CLINICAL TRIAL: NCT01525186
Title: The Relationship of Parental Feeding Control Practices to Food Intake of 3-5Yr Children in Families With Limited Incomes
Brief Title: Observational Study of Parental Feeding Practices to Improve Child's Food Intake and Weight Status
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Sponsor
Other Study IDs: MSUIRB 09-451
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Obesity; Feeding Behaviors
Keywords: Weight; Food intakes; Feeding
MeSH Terms: conditions — Obesity; Feeding Behavior; Body Weight

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background:

A topic of interest in the etiology of child obesity is if and how parental feeding behaviors are associated with child food intake and weight status.

Objectives:

The objective was to explore if and how directive (overt) and non-directive (covert and food environmental structure) types of parental feeding control were associated with children's food intake and weight status.

Design:

This was a cross-sectional, exploratory study using structural equation modeling to determine directional associations between maternal feeding practices and their child's food intakes and weight status. Researchers collected data from 330 dyads of 3-5yr children and mothers participating in a federal preschool program for low-income families (Head Start) in Michigan. Mothers' feeding practices (directive and non-directive control), children's food intakes, height and weight of both mothers and children were measured. Structural equation models tested the relationships between maternal feeding practices, the child's food intake and weight status.

Hypotheses:

1. Child weight is negatively associated with parents' directive feeding control practices.
2. Less directive control or greater non-directive control is associated with healthier food intakes in children.

ELIGIBILITY:
Inclusion Criteria:

* Dyads of child (3-5yrs) and the primary female caregiver
* Participating Head Start program in central Michigan

Exclusion Criteria:

* Children with disability except speech disorders
* Caregivers younger than 18 years old

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Low income mother and preschool children participating national school readiness program, HeadStart.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hoerr, PhD, Principal Investigator — Michigan State University

REFERENCES:
- [Derived] Murashima M, Hoerr SL, Hughes SO, Kaplowitz SA. Feeding behaviors of low-income mothers: directive control relates to a lower BMI in children, and a nondirective control relates to a healthier diet in preschoolers. Am J Clin Nutr. 2012 May;95(5):1031-7. doi: 10.3945/ajcn.111.024257. Epub 2012 Mar 28. PMID 22456658